CLINICAL TRIAL: NCT00624650
Title: Hemodynamics and Extravascular Lung Water in Acute Lung Injury: A Prospective Randomized Controlled Multicentered Trial of Goal Directed Treatment of EVLW Versus Standard Management for the Treatment of Acute Lung Injury
Brief Title: Hemodynamics and Extravascular Lung Water in Acute Lung Injury
Acronym: HEAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Pulsion Medical Systems (Industry); Oregon Clinical and Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00003491; IRB #e2978
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Acute Lung Injury
Keywords: Acute Lung Injury; Extravascular Lung Water; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome | interventions — Diuresis; Furosemide; Crystalloid Solutions; Albumins; Vasoconstrictor Agents; Norepinephrine; Vasopressins; Phenylephrine; Epinephrine; Dobutamine; Nutritional Status; Dialysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified FACTT (control) (Active Comparator): The investigators control arm consists of a simplified algorithm for conservative management of fluids in patients with ALI, as to be published by the ARDSnet group, based on the protocol used in the FACTT trial. The protocol calls for strict adherence to ARDSnet ventilation, our weaning protocol and use of only select vasoactive, beta-adrenergic drugs as it is felt that variation in these treatments could seriously confound our results. Albuterol administration will not be permitted in the either arm except for life threatening bronchospasm not responsive to ipratropium. Ipratropium may be administered at the treating physician's discretion for bronchospasm. PiCCO's will be placed in each control patient and data recorded twice daily. The treating physician's will be blinded to this data.
  Interventions: Drug: Diuresis (furosemide) part I; Other: Fluid Bolus (crystalloid or albumin); Drug: Vasopressors (Norepinephrine, Vasopressin, Phenylephrine, Epinephrine); Drug: Dobutamine; Drug: Diuresis (furosemide) part II; Procedure: Dialysis
- EVLW (Experimental): When EVLW exceeds 9 ml/kg PBW the algorithmic treatment is begun and continued until EVLW ≤9 ml/kg PBW or extubation whichever comes first as tolerated (see figure 6). Furosemide and volume contraction are initiated when sufficient volumetric preload (GEDI) is available to enact volume contraction as a means to decrease measured EVLW without causing concomitant hypoperfusion. Fluid administration is also guided by changes in EVLW. An increase in EVLW > 2ml/kg PBW as a result of fluid administration curtails any further fluid administration until the next scheduled measurement.
  Our ultimate treatment goal is to maximally lower EVLW towards the normal range - thus improving lung mechanics and gas exchange - without causing concomitant hemodynamic compromise and end-organ injury. By doing so we feel this algorithmic, goal directed, therapeutic approach should improve outcome.
  Interventions: Drug: Diuresis (furosemide) part I; Other: Fluid Bolus (crystalloid or albumin); Drug: Vasopressors (Norepinephrine, Vasopressin, Phenylephrine, Epinephrine); Drug: Dobutamine; Other: Concentrate all drips and nutrition; Drug: Diuresis (furosemide) part II; Procedure: Dialysis

INTERVENTIONS:
Drug: Diuresis (furosemide) part I — Goal: Overall I/O net negative 50ml/hour
  Initiation:
  1. Continuous IV furosemide at 3mg/hour or last known protocol specified dose
  2. Titrate up or down by 3mg/hour increments every hour as needed to establish diuresis goal
  3. Do not exceed 30mg/hour
  Furosemide Bolus:
  1. If unable to establish adequate diuresis at maximum dose may attempt furosemide bolusing as follows
  2. By intravenous bolus give 30, then 60, then 80, and 120 mg - one bolus dose every hour until urine output results in 1 ml/kg PBW/hr net negative fluid balance per hour
  3. Bolusing trials may be done at will but total furosemide dose may not exceed 800mg/24hour period
Other: Fluid Bolus (crystalloid or albumin) — 15 ml/kg PBW crystalloid (round to nearest 250 ml) or 25 grams albumin as rapidly as possible. Used for patients with a measured CVP<8 or measured PaOP <12mmHg in addition to concurrent urine output of <0.5 ml/kg/hr
  Arms: Modified FACTT (control)
Other: Fluid Bolus (crystalloid or albumin) — 10 ml/kg PBW crystalloid (round to nearest 70ml) or 25 grams albumin as rapidly as possible.
  Perform thermodilution immediately before and after and 60 minutes after each bolus. If EVLW increases > 2ml/kg PBW within 60 minutes after a bolus do not give any further boluses until next regularly scheduled measurement. This therapy is available for patients with a map < 60 or who are on vasopressors that also have a measured GEDI less than goal
  Arms: EVLW
Drug: Vasopressors (Norepinephrine, Vasopressin, Phenylephrine, Epinephrine) — (may use any alone or in combination)
  1. Norepinephrine - 0.05mcg/kg/min - increase for effect not to exceed (NTE) 1mcg/kg/min.
  2. Vasopressin - 0.04 international units/hour
  3. Phenylephrine - 7mcg/min - may increase to for effect not to exceed 500mcg/min.
  4. Epinephrine - 1 mcg/min - may increase for effect not to exceed 20mcg/min.
  Weaning: When MAP ≥ 60 mm/Hg on stable dose of vasopressor begin reduction of vasopressor by greater than or equal to 25% stabilizing dose at intervals ≤ 4 hours to maintain MAP ≥ 60 mm/Hg.
  Arms: Modified FACTT (control)
Drug: Vasopressors (Norepinephrine, Vasopressin, Phenylephrine, Epinephrine) — (may use alone or in combination)
  1. Norepinephrine - 0.05mcg/kg/min - increase for effect not to exceed (NTE) 1mcg/kg/min.
  2. Vasopressin - 0.04 international units/hour
  3. Phenylephrine - 7mcg/min - may increase to for effect not to exceed 500mcg/min.
  4. Epinephrine - 1 mcg/min - may increase for effect not to exceed 20mcg/min.
  Weaning: When MAP ≥ 60 mm/Hg on stable dose of vasopressor begin reduction of vasopressor by greater than or equal to 25% stabilizing dose at intervals ≤ 4 hours to maintain MAP ≥ 60 mm/Hg.
  In the experimental arm vasopressors are a treatment option in patients with a Mean Arterial Pressure of < 60
  Arms: EVLW
Drug: Dobutamine — 1. Begin at 5mcg/kg/min and increase by 3 mcg/kg/min increments at 15 minute intervals until C.I. ≥ 2.5 or maximum dose of 20mcg/kg/min has been reached.
  2. Begin weaning 4 hours after low CI is reversed. Wean by ≥ 25% of the stabilizing dose at intervals of ≤ 4 hours to maintain hemodynamic algorithm goals.
  3. If patient is on dobutamine as a result of an earlier cell assignment, dobutamine should be ignored for the purpose of subsequent assignment, but should be continued to be weaned per protocol.
  Used in patients with a measured cardiac index < 2.5
  Arms: EVLW
Drug: Dobutamine — 1. Begin at 5mcg/kg/min and increase by 3 mcg/kg/min increments at 15 minute intervals until C.I. ≥ 2.5 or maximum dose of 20mcg/kg/min has been reached.
  2. Begin weaning 4 hours after low CI is reversed. Wean by ≥ 25% of the stabilizing dose at intervals of ≤ 4 hours to maintain hemodynamic algorithm goals.
  3. If patient is on dobutamine as a result of an earlier cell assignment, dobutamine should be ignored for the purpose of subsequent assignment, but should be continued to be weaned per protocol.
  Arms: Modified FACTT (control)
Other: Concentrate all drips and nutrition — Concentrate all drips and nutrition in order to minimize fluid volume as much as possible. Intravenous fluid to be run at keep vein open rate.
  EVLW arm: Patients with a MAP > 60 and off vasopressors for >12 hours, as well as patients with a measured cardiac index >2.5 that also have a measured GEDI > goal.
  Arms: EVLW
Drug: Diuresis (furosemide) part II — Withhold furosemide if:
  1. Significant hypokalemia (K+ <= 2.5 meq/L), or hypernatremia (Na+ >= 155 meq/L) occurs within last 12 hours may then be restarted if the prevailing condition no longer exists
  2. Dialysis dependence
  3. Oliguria (less than 0.5ml/kg/hour) with either creatinine > 3, or clinical suspicion of rapidly evolving ARF
  4. More than 800mg has been given in less then 24 hours
  5. Creatinine increases > 1.5 mg/dl in any 24 hour period
Procedure: Dialysis — 1. Need for CVVHD or intermittent hemodialysis to be determined by treating clinicians.
  2. CVC arm: If fluid management to be accomplished with dialysis then fluid balance goals to be determined per clinicians.
  3. EVLW arm: Fluid balance as per algorithm
  4. When using intermittent HD it is recommended that no more than 2 liters net negative fluid is removed per dialysis session. Total fluid removal per run to be estimated by the clinicians to attain CVP or GEDI goals per algorithm.

SUMMARY:
The purpose of this study is to test a treatment that tries to reduce the amount of fluid in the lungs of subjects with acute lung injury to see if this is helpful.

DETAILED DESCRIPTION:
The objective of this study is to conduct a randomized, controlled trial of a goal directed therapy designed to improve outcome in patients with acute lung injury (ALI). The investigators are comparing two algorithmic approaches in managing patients with ALI - one, the control arm, attempts to reduce the amount of fluid in the lung in patients with ALI by diuresis based on central venous pressure and urine output, the other the treatment arm attempting to reduce lung water by directing therapy to measured lung water and using more sensitive indicators of preload status than CVP. The protocol uses measured extravascular lung water (EVLW) to direct diuresis and appropriate fluid restriction in a goal directed fashion in order to lower EVLW towards the normal range.

ELIGIBILITY:
Inclusion Criteria:

Acute onset of:

1. PaO2/FiO2 less than or equal to 300.
2. Bilateral infiltrates consistent with pulmonary edema on the frontal chest radiograph.
3. Requirement for positive pressure ventilation through an endotracheal tube or tracheostomy.
4. No clinical evidence of left atrial hypertension that would explain the pulmonary infiltrates. If measured, pulmonary arterial wedge pressure less than or equal to 18 mmHg.

Exclusion Criteria:

1. Age younger than 18 years old.
2. Greater than 24 hours since all inclusion criteria first met.
3. Neuromuscular disease that impairs ability to ventilate without assistance, such as C5 or higher spinal cord injury, amyotrophic lateral sclerosis, Guillain-Barré syndrome, myasthenia gravis, or kyphoscoliosis (see Appendix I.A).
4. Pregnancy (negative pregnancy test required for women of child-bearing potential).
5. Severe chronic respiratory disease (see Appendix I.C).
6. Severe Chronic Liver Disease (Child-Pugh 11 - 15, see Appendix I.E)
7. Weight > 160 kg.
8. Burns greater than 70% total body surface area.
9. Malignancy or other irreversible disease or conditions for which 6-month mortality is estimated to be greater than 50 % (see Appendix I.A).
10. Known cardiac or vascular aneurysm.
11. Contraindications to femoral arterial puncture - platelets < 30, bilateral femoral arterial grafts, INR > 3.0.
12. Not committed to full support.
13. Participation in other experimental medication trial within 30 days.
14. Allergy to intravenous lasix or any components of its carrier.
15. History of severe CHF - NYHA class ≥ III, previously documented EF < 30%.
16. Diffuse alveolar hemorrhage.
17. Presence of reactive airway disease (active will be defined based on recent frequency and amounts of MDI's use and steroids to control the disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Phillips, M.D., Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Kaiser Permanente Sunnyside, Clackamas, Oregon
  - Legacy Good Samaritan, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon

REFERENCES:
- [Background] Ware LB, Matthay MA. The acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1334-49. doi: 10.1056/NEJM200005043421806. No abstract available. PMID 10793167
- [Background] Matthay MA. Alveolar fluid clearance in patients with ARDS: does it make a difference? Chest. 2002 Dec;122(6 Suppl):340S-343S. doi: 10.1378/chest.122.6_suppl.340s. PMID 12475812
- [Background] Mitchell JP, Schuller D, Calandrino FS, Schuster DP. Improved outcome based on fluid management in critically ill patients requiring pulmonary artery catheterization. Am Rev Respir Dis. 1992 May;145(5):990-8. doi: 10.1164/ajrccm/145.5.990. PMID 1586077
- [Background] Eisenberg PR, Hansbrough JR, Anderson D, Schuster DP. A prospective study of lung water measurements during patient management in an intensive care unit. Am Rev Respir Dis. 1987 Sep;136(3):662-8. doi: 10.1164/ajrccm/136.3.662. PMID 3307570
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Bendjelid K, Romand JA. Fluid responsiveness in mechanically ventilated patients: a review of indices used in intensive care. Intensive Care Med. 2003 Mar;29(3):352-60. doi: 10.1007/s00134-002-1615-9. Epub 2003 Jan 21. PMID 12536268
- [Background] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Background] Goedje O, Seebauer T, Peyerl M, Pfeiffer UJ, Reichart B. Hemodynamic monitoring by double-indicator dilution technique in patients after orthotopic heart transplantation. Chest. 2000 Sep;118(3):775-81. doi: 10.1378/chest.118.3.775. PMID 10988202
- [Background] Bernard GR. Acute respiratory distress syndrome: a historical perspective. Am J Respir Crit Care Med. 2005 Oct 1;172(7):798-806. doi: 10.1164/rccm.200504-663OE. Epub 2005 Jul 14. PMID 16020801
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Background] Matthay MA, Zimmerman GA. Acute lung injury and the acute respiratory distress syndrome: four decades of inquiry into pathogenesis and rational management. Am J Respir Cell Mol Biol. 2005 Oct;33(4):319-27. doi: 10.1165/rcmb.F305. No abstract available. PMID 16172252
- [Background] Groeneveld AB, Polderman KH. Acute lung injury, overhydration or both? Crit Care. 2005 Apr;9(2):136-7. doi: 10.1186/cc3039. Epub 2005 Jan 17. PMID 15774062
- [Background] Ware LB, Matthay MA. Alveolar fluid clearance is impaired in the majority of patients with acute lung injury and the acute respiratory distress syndrome. Am J Respir Crit Care Med. 2001 May;163(6):1376-83. doi: 10.1164/ajrccm.163.6.2004035. PMID 11371404
- [Background] Sakka SG, Klein M, Reinhart K, Meier-Hellmann A. Prognostic value of extravascular lung water in critically ill patients. Chest. 2002 Dec;122(6):2080-6. doi: 10.1378/chest.122.6.2080. PMID 12475851
- [Background] Phillips, C.R., Smith S. Extravascular Lung Water In Early ARDS ATS Poster Exhibit, 2006
- [Background] Sartori C, Matthay MA. Alveolar epithelial fluid transport in acute lung injury: new insights. Eur Respir J. 2002 Nov;20(5):1299-313. doi: 10.1183/09031936.02.00401602. PMID 12449188
- [Background] Sporn P. Keep the lung dry--sense or nonsense? Acta Anaesthesiol Scand Suppl. 1996;109:63-5. No abstract available. PMID 8901949
- [Background] Martin GS, Eaton S, Mealer M, Moss M. Extravascular lung water in patients with severe sepsis: a prospective cohort study. Crit Care. 2005 Apr;9(2):R74-82. doi: 10.1186/cc3025. Epub 2005 Jan 11. PMID 15774053
- [Background] Martin GS, Moss M, Wheeler AP, Mealer M, Morris JA, Bernard GR. A randomized, controlled trial of furosemide with or without albumin in hypoproteinemic patients with acute lung injury. Crit Care Med. 2005 Aug;33(8):1681-7. doi: 10.1097/01.ccm.0000171539.47006.02. PMID 16096441
- [Background] Perkins GD, McAuley DF, Thickett DR, Gao F. The beta-agonist lung injury trial (BALTI): a randomized placebo-controlled clinical trial. Am J Respir Crit Care Med. 2006 Feb 1;173(3):281-7. doi: 10.1164/rccm.200508-1302OC. Epub 2005 Oct 27. PMID 16254268
- [Background] Elings VB, Lewis FR. A single indicator technique to estimate extravascular lung water. J Surg Res. 1982 Nov;33(5):375-85. doi: 10.1016/0022-4804(82)90052-x. PMID 6752580
- [Background] Mihm FG, Feeley TW, Rosenthal MH, Lewis F. Measurement of extravascular lung water in dogs using the thermal-green dye indicator dilution method. Anesthesiology. 1982 Aug;57(2):116-22. doi: 10.1097/00000542-198208000-00009. PMID 7046519
- [Background] Mihm FG, Feeley TW, Jamieson SW. Thermal dye double indicator dilution measurement of lung water in man: comparison with gravimetric measurements. Thorax. 1987 Jan;42(1):72-6. doi: 10.1136/thx.42.1.72. PMID 3616974
- [Background] Sivak ED, Tita J, Meden G, Ishigami M, Graves J, Kavlich J, Stowe NT, Magnusson MO. Effects of furosemide versus isolated ultrafiltration on extravascular lung water in oleic acid-induced pulmonary edema. Crit Care Med. 1986 Jan;14(1):48-51. doi: 10.1097/00003246-198601000-00011. PMID 3940754
- [Background] Wickerts CJ, Blomqvist H, Berg B, Rosblad PG, Hedenstierna G. Furosemide, when used in combination with positive end-expiratory pressure, facilitates the resorption of extravascular lung water in experimental hydrostatic pulmonary oedema. Acta Anaesthesiol Scand. 1991 Nov;35(8):776-83. doi: 10.1111/j.1399-6576.1991.tb03390.x. PMID 1763601
- [Background] Waugh JB, Op't Holt TB, Gadek JE, Clanton TL. High-dose furosemide alters gas exchange in a model of acute lung injury. J Crit Care. 1996 Sep;11(3):129-37. doi: 10.1016/s0883-9441(96)90009-x. PMID 8891964
- [Background] Reising CA, Chendrasekhar A, Wall PL, Paradise NF, Timberlake GA, Moorman DW. Continuous dose furosemide as a therapeutic approach to acute respiratory distress syndrome (ARDS). J Surg Res. 1999 Mar;82(1):56-60. doi: 10.1006/jsre.1998.5513. PMID 10068526
- [Background] Martin GS. Fluid balance and colloid osmotic pressure in acute respiratory failure: emerging clinical evidence. Crit Care. 2000;4 Suppl 2(Suppl 2):S21-5. doi: 10.1186/cc966. Epub 2000 Oct 13. PMID 11255595
- [Background] Martin GS, Mangialardi RJ, Wheeler AP, Dupont WD, Morris JA, Bernard GR. Albumin and furosemide therapy in hypoproteinemic patients with acute lung injury. Crit Care Med. 2002 Oct;30(10):2175-82. doi: 10.1097/00003246-200210000-00001. PMID 12394941
- [Background] Mojtahedzadeh M, Vazin A, Najafi A, Khalilzadeh A, Abdollahi M. The effect of furosemide infusion on serum epidermal growth factor concentration after acute lung injury. J Infus Nurs. 2005 May-Jun;28(3):188-93. doi: 10.1097/00129804-200505000-00007. PMID 15912074
- [Background] Molloy WD, Lee KY, Girling L, Prewitt RM. Treatment of canine permeability pulmonary edema: short-term effects of dobutamine, furosemide, and hydralazine. Circulation. 1985 Dec;72(6):1365-71. doi: 10.1161/01.cir.72.6.1365. PMID 4064278
- [Background] Ali J, Wood LD. Pulmonary vascular effects of furosemide on gas exchange in pulmonary edema. J Appl Physiol Respir Environ Exerc Physiol. 1984 Jul;57(1):160-7. doi: 10.1152/jappl.1984.57.1.160. PMID 6469777
- [Background] Ali J, Unruh H, Skoog C, Goldberg HS. The effect of lung edema on pulmonary vasoactivity of furosemide. J Surg Res. 1983 Nov;35(5):383-90. doi: 10.1016/0022-4804(83)90027-6. PMID 6632865
- [Background] Ali J, Chernicki W, Wood LD. Effect of furosemide in canine low-pressure pulmonary edema. J Clin Invest. 1979 Nov;64(5):1494-504. doi: 10.1172/JCI109608. PMID 500821
- [Background] Hechtman HB, Weisel RD, Vito L, Ali J, Berger RL. The independence of pulmonary shunting and pulmonary edema. Surgery. 1973 Aug;74(2):300-6. No abstract available. PMID 4577807
- [Background] Baltopoulos G, Zakynthinos S, Dimopoulos A, Roussos C. Effects of furosemide on pulmonary shunts. Chest. 1989 Sep;96(3):494-8. doi: 10.1378/chest.96.3.494. PMID 2670464
- [Background] Boussat S, Jacques T, Levy B, Laurent E, Gache A, Capellier G, Neidhardt A. Intravascular volume monitoring and extravascular lung water in septic patients with pulmonary edema. Intensive Care Med. 2002 Jun;28(6):712-8. doi: 10.1007/s00134-002-1286-6. Epub 2002 May 18. PMID 12107676
- [Background] Halperin BD, Feeley TW, Mihm FG, Chiles C, Guthaner DF, Blank NE. Evaluation of the portable chest roentgenogram for quantitating extravascular lung water in critically ill adults. Chest. 1985 Nov;88(5):649-52. doi: 10.1378/chest.88.5.649. PMID 3902385
- [Background] Meade MO, Cook RJ, Guyatt GH, Groll R, Kachura JR, Bedard M, Cook DJ, Slutsky AS, Stewart TE. Interobserver variation in interpreting chest radiographs for the diagnosis of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2000 Jan;161(1):85-90. doi: 10.1164/ajrccm.161.1.9809003. PMID 10619802
- [Background] Baudendistel L, Shields JB, Kaminski DL. Comparison of double indicator thermodilution measurements of extravascular lung water (EVLW) with radiographic estimation of lung water in trauma patients. J Trauma. 1982 Dec;22(12):983-8. doi: 10.1097/00005373-198212000-00002. PMID 7143511
- [Background] Roch A, Michelet P, Lambert D, Delliaux S, Saby C, Perrin G, Ghez O, Bregeon F, Thomas P, Carpentier JP, Papazian L, Auffray JP. Accuracy of the double indicator method for measurement of extravascular lung water depends on the type of acute lung injury. Crit Care Med. 2004 Mar;32(3):811-7. doi: 10.1097/01.ccm.0000114831.59185.02. PMID 15090967
- [Background] Kirov MY, Kuzkov VV, Kuklin VN, Waerhaug K, Bjertnaes LJ. Extravascular lung water assessed by transpulmonary single thermodilution and postmortem gravimetry in sheep. Crit Care. 2004 Dec;8(6):R451-8. doi: 10.1186/cc2974. Epub 2004 Oct 19. PMID 15566591
- [Background] Rossi P, Oldner A, Wanecek M, Leksell LG, Rudehill A, Konrad D, Weitzberg E. Comparison of gravimetric and a double-indicator dilution technique for assessment of extra-vascular lung water in endotoxaemia. Intensive Care Med. 2003 Mar;29(3):460-6. doi: 10.1007/s00134-002-1604-z. Epub 2003 Feb 8. PMID 12577158
- [Background] Katzenelson R, Perel A, Berkenstadt H, Preisman S, Kogan S, Sternik L, Segal E. Accuracy of transpulmonary thermodilution versus gravimetric measurement of extravascular lung water. Crit Care Med. 2004 Jul;32(7):1550-4. doi: 10.1097/01.ccm.0000130995.18334.8b. PMID 15241101
- [Background] Fernandez-Mondejar E, Rivera-Fernandez R, Garcia-Delgado M, Touma A, Machado J, Chavero J. Small increases in extravascular lung water are accurately detected by transpulmonary thermodilution. J Trauma. 2005 Dec;59(6):1420-3; discussion 1424. doi: 10.1097/01.ta.0000198360.01080.42. PMID 16394916
- [Background] Nuckton TJ, Alonso JA, Kallet RH, Daniel BM, Pittet JF, Eisner MD, Matthay MA. Pulmonary dead-space fraction as a risk factor for death in the acute respiratory distress syndrome. N Engl J Med. 2002 Apr 25;346(17):1281-6. doi: 10.1056/NEJMoa012835. PMID 11973365
- [Background] Tavernier B, Makhotine O, Lebuffe G, Dupont J, Scherpereel P. Systolic pressure variation as a guide to fluid therapy in patients with sepsis-induced hypotension. Anesthesiology. 1998 Dec;89(6):1313-21. doi: 10.1097/00000542-199812000-00007. PMID 9856704
- [Background] Calvin JE, Driedger AA, Sibbald WJ. The hemodynamic effect of rapid fluid infusion in critically ill patients. Surgery. 1981 Jul;90(1):61-76. PMID 7245052
- [Background] Schneider AJ, Teule GJ, Groeneveld AB, Nauta J, Heidendal GA, Thijs LG. Biventricular performance during volume loading in patients with early septic shock, with emphasis on the right ventricle: a combined hemodynamic and radionuclide study. Am Heart J. 1988 Jul;116(1 Pt 1):103-12. doi: 10.1016/0002-8703(88)90256-6. PMID 3394612
- [Background] Reuse C, Vincent JL, Pinsky MR. Measurements of right ventricular volumes during fluid challenge. Chest. 1990 Dec;98(6):1450-4. doi: 10.1378/chest.98.6.1450. PMID 2245688
- [Background] Wagner JG, Leatherman JW. Right ventricular end-diastolic volume as a predictor of the hemodynamic response to a fluid challenge. Chest. 1998 Apr;113(4):1048-54. doi: 10.1378/chest.113.4.1048. PMID 9554646
- [Background] Magder S, Lagonidis D. Effectiveness of albumin versus normal saline as a test of volume responsiveness in post-cardiac surgery patients. J Crit Care. 1999 Dec;14(4):164-71. doi: 10.1016/s0883-9441(99)90030-8. PMID 10622750
- [Background] Tousignant CP, Walsh F, Mazer CD. The use of transesophageal echocardiography for preload assessment in critically ill patients. Anesth Analg. 2000 Feb;90(2):351-5. doi: 10.1097/00000539-200002000-00021. PMID 10648320
- [Background] Michard F, Boussat S, Chemla D, Anguel N, Mercat A, Lecarpentier Y, Richard C, Pinsky MR, Teboul JL. Relation between respiratory changes in arterial pulse pressure and fluid responsiveness in septic patients with acute circulatory failure. Am J Respir Crit Care Med. 2000 Jul;162(1):134-8. doi: 10.1164/ajrccm.162.1.9903035. PMID 10903232
- [Background] Feissel M, Michard F, Mangin I, Ruyer O, Faller JP, Teboul JL. Respiratory changes in aortic blood velocity as an indicator of fluid responsiveness in ventilated patients with septic shock. Chest. 2001 Mar;119(3):867-73. doi: 10.1378/chest.119.3.867. PMID 11243970
- [Background] Martin GS, Ely EW, Carroll FE, Bernard GR. Findings on the portable chest radiograph correlate with fluid balance in critically ill patients. Chest. 2002 Dec;122(6):2087-95. doi: 10.1378/chest.122.6.2087. PMID 12475852
- [Background] Ely EW, Smith AC, Chiles C, Aquino SL, Harle TS, Evans GW, Haponik EF. Radiologic determination of intravascular volume status using portable, digital chest radiography: a prospective investigation in 100 patients. Crit Care Med. 2001 Aug;29(8):1502-12. doi: 10.1097/00003246-200108000-00002. PMID 11505116
- [Background] Michard F. Underutilized tools for the assessment of intravascular volume status. Chest. 2003 Jul;124(1):414-5; author reply 415-6. No abstract available. PMID 12853559
- [Background] Connors AF Jr. The role of right heart catheterization in the care of the critically ill: benefits, limitations, and risks. Int J Cardiol. 1983 Nov-Dec;4(4):474-7. doi: 10.1016/0167-5273(83)90200-0. No abstract available. PMID 6642783
- [Background] Diebel LN, Wilson RF, Tagett MG, Kline RA. End-diastolic volume. A better indicator of preload in the critically ill. Arch Surg. 1992 Jul;127(7):817-21; discussion 821-2. doi: 10.1001/archsurg.1992.01420070081015. PMID 1524482
- [Background] Tomicic V, Graf J, Echevarria G, Espinoza M, Abarca J, Montes JM, Torres J, Nunez G, Guerrero J, Luppi M, Canals C. [Intrathoracic blood volume versus pulmonary artery occlusion pressure as estimators of cardiac preload in critically ill patients]. Rev Med Chil. 2005 Jun;133(6):625-31. doi: 10.4067/s0034-98872005000600001. Epub 2005 Jul 22. Spanish. PMID 16075124
- [Background] Szakmany T, Toth I, Kovacs Z, Leiner T, Mikor A, Koszegi T, Molnar Z. Effects of volumetric vs. pressure-guided fluid therapy on postoperative inflammatory response: a prospective, randomized clinical trial. Intensive Care Med. 2005 May;31(5):656-63. doi: 10.1007/s00134-005-2606-4. Epub 2005 Apr 6. PMID 15812629
- [Background] Nirmalan M, Willard TM, Edwards DJ, Little RA, Dark PM. Estimation of errors in determining intrathoracic blood volume using the single transpulmonary thermal dilution technique in hypovolemic shock. Anesthesiology. 2005 Oct;103(4):805-12. doi: 10.1097/00000542-200510000-00019. PMID 16192773
- [Background] Hofmann D, Klein M, Wegscheider K, Sakka SG. [Extended hemodynamic monitoring using transpulmonary thermodilution Influence of various factors on the accuracy of the estimation of intrathoracic blood volume and extravascular lung water in critically ill patients]. Anaesthesist. 2005 Apr;54(4):319-26. doi: 10.1007/s00101-005-0809-2. German. PMID 15726244
- [Background] Donati A, Loggi S, Coltrinari R, Pelaia P. Intrathoracic blood volume as index of cardiac output variations. Acta Anaesthesiol Scand. 2004 Mar;48(3):386-7. doi: 10.1111/j.0001-5172.2004.0320c.x. No abstract available. PMID 14982579
- [Background] Sakka SG, Meier-Hellmann A. Intrathoracic blood volume in a patient with pulmonary embolism. Eur J Anaesthesiol. 2003 Mar;20(3):256-7. doi: 10.1017/s0265021503230428. No abstract available. PMID 12650499
- [Background] Kuz'kov VV, Kirov MIu, Nedashkovskii EV. [Volumetric monitoring based on transpulmonary thermodilution in anesthesiology and intensive care]. Anesteziol Reanimatol. 2003 Jul-Aug;(4):67-73. Russian. PMID 14524028
- [Background] Reuter DA, Felbinger TW, Moerstedt K, Weis F, Schmidt C, Kilger E, Goetz AE. Intrathoracic blood volume index measured by thermodilution for preload monitoring after cardiac surgery. J Cardiothorac Vasc Anesth. 2002 Apr;16(2):191-5. doi: 10.1053/jcan.2002.31064. PMID 11957169
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Eisner MD, Thompson T, Hudson LD, Luce JM, Hayden D, Schoenfeld D, Matthay MA; Acute Respiratory Distress Syndrome Network. Efficacy of low tidal volume ventilation in patients with different clinical risk factors for acute lung injury and the acute respiratory distress syndrome. Am J Respir Crit Care Med. 2001 Jul 15;164(2):231-6. doi: 10.1164/ajrccm.164.2.2011093. PMID 11463593
- [Background] Doyle RL, Szaflarski N, Modin GW, Wiener-Kronish JP, Matthay MA. Identification of patients with acute lung injury. Predictors of mortality. Am J Respir Crit Care Med. 1995 Dec;152(6 Pt 1):1818-24. doi: 10.1164/ajrccm.152.6.8520742.
- [Background] Frezza EE, Mezghebe H. Indications and complications of arterial catheter use in surgical or medical intensive care units: analysis of 4932 patients. Am Surg. 1998 Feb;64(2):127-31. PMID 9486883
- [Background] Dorman T, Breslow MJ, Lipsett PA, Rosenberg JM, Balser JR, Almog Y, Rosenfeld BA. Radial artery pressure monitoring underestimates central arterial pressure during vasopressor therapy in critically ill surgical patients. Crit Care Med. 1998 Oct;26(10):1646-9. doi: 10.1097/00003246-199810000-00014. PMID 9781720
- [Background] MacIntyre NR. Current issues in mechanical ventilation for respiratory failure. Chest. 2005 Nov;128(5 Suppl 2):561S-567S. doi: 10.1378/chest.128.5_suppl_2.561S. PMID 16306054
- [Background] Steinberg KP, Mitchell DR, Maunder RJ, Milberg JA, Whitcomb ME, Hudson LD. Safety of bronchoalveolar lavage in patients with adult respiratory distress syndrome. Am Rev Respir Dis. 1993 Sep;148(3):556-61. doi: 10.1164/ajrccm/148.3.556. PMID 8368623
- [Background] Brown DL, Hungness ES, Campbell RS, Luchette FA. Ventilator-associated pneumonia in the surgical intensive care unit. J Trauma. 2001 Dec;51(6):1207-16. doi: 10.1097/00005373-200112000-00034. No abstract available. PMID 11740281
- [Background] Rouby JJ, Martin De Lassale E, Poete P, Nicolas MH, Bodin L, Jarlier V, Le Charpentier Y, Grosset J, Viars P. Nosocomial bronchopneumonia in the critically ill. Histologic and bacteriologic aspects. Am Rev Respir Dis. 1992 Oct;146(4):1059-66. doi: 10.1164/ajrccm/146.4.1059. PMID 1416397
- [Background] Chesnutt AN, Matthay MA, Tibayan FA, Clark JG. Early detection of type III procollagen peptide in acute lung injury. Pathogenetic and prognostic significance. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):840-5. doi: 10.1164/ajrccm.156.3.9701124. PMID 9310002

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Modified FACTT (Control) | EVLW
Started | 17 | 16
Completed | 16 | 15
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified FACTT (Control) | EVLW | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 4 | 10 | 14
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Variable Will be the Total Reduction in Measured Lung Water
Time Frame: The first seven days of treatment
Population: The study's Principal Investigator departed the institution before analyses were conducted. OHSU will never have analyses complete for this study. The study device is no longer manufactured.
Arm/Group | Modified FACTT (Control) | EVLW
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Modified FACTT (Control) | EVLW
All-Cause Mortality (participants affected / at risk) | 2/17 | 5/16
Serious Adverse Events (participants affected / at risk) | 2/17 | 5/16
Other Adverse Events (participants affected / at risk) | 1/17 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modified FACTT (Control) (N=17) | EVLW (N=16)
Death (Cardiac disorders) | 2 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Modified FACTT (Control) (N=17) | EVLW (N=16)
Hypernatremia (Renal and urinary disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Principal Investigator departed the institution before Primary Outcome Measure analyses were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No